CLINICAL TRIAL: NCT00592618
Title: Effect of NAC on Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 346147SLEEP
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2007-05

CONDITIONS: ESRD; Sleep Apnea
Keywords: ESRD; Hemodialysis; Sleep Apnea
MeSH Terms: conditions — Kidney Failure, Chronic; Sleep Apnea Syndromes | interventions — Acetylcysteine

INTERVENTIONS:
Drug: Oral N-Acetylcysteine 1200 mg x 2/day for 4 weeks

SUMMARY:
Sleep studies in ESRD patients have identified increased prevalence of Sleep Apnea. Based on current knowledge, treatment aimed at reducing oxidative stress might improve Sleep Apnea in HD patients. The aim of our study is to investigate the effect of N-acetylsysteine on Sleep Apnea in HD patients.

DETAILED DESCRIPTION:
Background Cardiovascular disease is the commonest cause of morbidity and mortality in chronic dialysis patients [1]. Sleep studies in ESRD patients have identified increased prevalence of sleep apnea (SA), both obstructive (OSA) and central (CSA) in origin [2]. The reported prevalence of SA in patients with ESRD ranges from 50% to 70% [3], which is dramatically higher than the estimated prevalence of 2% to 4% in the general population [4]. SA has been recognized as a novel risk factor for cardiovascular disease in general population [5]. Recent evidence showed that severity of SA in hemodialysis patients is associated with severity of coronary artery calcifications [6]. Underlying mechanisms by which SA adversely affects cardiovascular morbidity and mortality have not been fully established yet. The presence of untreated SA may further impair fluid balance, cardiovascular function and increase mortality through abnormal vagal or sympatomimetic responces and hypoxia [7]. One intriguing possibility is oxidative stress, which has been implicated in cardiovascular disease in patients with ESRD [8]. Recent study demonstrated association between SA and decreased antioxidant status in hemodialysis patients [6]. Repeated apnea-related hypoxic events in patients with SA may trigger elevated oxidative stress [9].

In general population, the treatment of SA with CPAP improves oxygenation during sleep and quality of life [10]. In the ESRD population, CPAP was used in a very preliminary study on 8 patients with some improvement in nocturnal oxygenation and 5 of 6 patients reported improved daytime alertness [11]. Unfortunately, CPAP application itself may be stressful, poorly tolerated and so disturb night sleep.

Hanly and Pierratos suggested that SA in hemodialysis patients may be a consequence of inadequate treatment of uremia by standard 4-hours thrice-weekly HD procedure [12]. This group reported that intensive nocturnal HD for 8 hours 6-7 times per week reduced the severity of SA, although their patients continued to suffer from frequent arousals, diminished sleep time, REM sleep and sleep efficiency [12]. Restoration of normal kidney function by transplantation may lead to reversal of SA [13, 14].

Several experimental and clinical studies showed that increased oxidative stress in dialysis patients may be due to inhibition of nitric oxide (NO) synthesis by ADMA (Asymmetric Dimethylarginine ), known to be endogenous inhibitor of NO synthetase [15]. ADMA may be significantly reduced by dialysis [16]. Metabolism of ADMA is primarily by the enzyme DDAH , which activity is decreased by inflammation, oxidative stress, diabetes mellitus and hypercholesterolemia [17 ]. It was proposed that circulating ADMA may be one mechanism accounting for the resistant hypertension and overfluid in dialysis patients [17 ].

Based on current knowledge, treatment aimed at reducing oxidative stress should decrease ADMA levels [17 ], and it is logical to suggest that such a therapy might improve SA in HD patients. One preliminary study on effect of antioxidant Vitamin E showed a small beneficial effect on ADMA in chronic kidney disease [19 ].

In our opinion, it is worth to check an ability of antioxidant therapy to produce a favorable effect on parameters of SA in dialysis patients.

N-Acetylcysteine (NAC) is an active antioxidant proved to be safe and beneficial in hemodialysis patents [19]. In our recent study, NAC effectively reduced the ototoxic effect of gentamicin in chronic hemodialysis patients [20, 21]. Cheap and safe drug therapy may appear more cost effective than such resource consuming therapies as CPAP and not readily available treatments as prolong every night hemodialysis or kidney transplantation.

The aim of our study is to investigate the effect of N-acetylsysteine on SA in HD patients.

Methods. Study population. The study will include 20 patients with ESRD, treated with chronic hemodialysis in Assaf Harofeh Medical Center and suffering from sleep disturbances, such as frequent arousals, snoring, daytime sleepiness.

Patients will be excluded from the study if they are:

1. Recently started treated with chronic dialysis: less than 3 months.
2. Survived recent major illness, requiring hospitalisation in the last 3 months.
3. Patients with acute renal failure
4. Currently treated with antioxidants ( NAC, vitamin E ets.)
5. Current use of sleep pills Study protocol. We planned this study as a prospective cross-sectional study where every patient will serve as his/her own control. Al the patients will continue their previous dialysis and drugs regimen. The presence and severity of SA will be accessed using the overnight polysomnography in the Sleep Laboratory.

After performance of baseline overnight polysomnography the patients will receive orally NAC 1200 mg x 2/day for 4 weeks. At the end of this therapy, a follow up overnight polysomnography examination will be performed.

The clinical monitoring of all the patients will include:

1. Blood Pressure and Heart Rate - at each dialysis session 3 times a week. .
2. Review of medications and doses.
3. Body weight - at each dialysis session 3 times a week
4. Dialysis adequacy: Kt/V at study start and end.
5. Biochemical studies: full chemistry, bicarbonate, ADMA, DDAH, NO - both at baseline and follow up visits.

Statistical analysis The statistical analysis will be performed using the statistical software SPSS-version 10. Parametric data will be expressed as means ± standard deviation and compared by the standard t-test. Non-parametric data will be compared using chi square test. p value of 0.05 or less will be considered significant.

References

1. United States Renal Data System. Patient mortality and survival. USRDS Annual Report. Am J Kidney Dis 1997; 30 [Suppl. 1]: s91-s101
2. Chakravorty I, Shastry M, Farrington K. Sleep apnoea in end-stage renal disease: a short review of mechanisms and potential benefit from its treatment. Nephrol Dial Transplant 2007; 22:28-31
3. Kraus M, Hamburger R. Sleep apnea in renal failure. Adv Perit Dial 1997; 13:88-92
4. Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults.

   NEJM 1993; 328:1230-35
5. Wolk R, Kara T, Somers V. Sleep-disordered breathing and cardiovascular disease.

   Circulation 2003;108:9-12
6. Jung H, Han H, Lee J. Sleep apnea, coronary artery disease, and antioxidant status in hemodialysis patients. AJKD 2005;45:875-882
7. Zoccali C. Sleep apnoea and nocturnal hypoxaemia in dialysis patients: mere risk-indicators or causal factors for cardiovascular disease? Nephrol Dial Transplant 2000, 15:1919-21
8. Boaz M, Matas Z, Biro A, Katzir Z, Green M, Fainaru M, Smetana S. Serum malondialdehyde and prevalent cardiovascular disease in hemodialysis. Kidney Int 1999;56:1078-83
9. Lavie L. Obstructive sleep apnoea syndrome--an oxidative stress disorder. Sleep Med Rev 2003;7:35-51
10. D'Ambrosio C, Bowman T, Mohsenin V. Quality of life in patients with obstructive sleep apnea: effect of nasal continuous positive airway pressure--a prospective study.Chest 1999;115:123-29
11. Pressman M, Benz R, Schleifer C, Peterson D. Sleep disordered breathing in ESRD: acute beneficial effects of treatment with nasal continuous positive airway pressure. Kidney Int 1993; 43:1134-39.
12. Hanly P, Pierratos A. Improvement of sleep apnea in patients with chronic renal failure who undergo nocturnal hemodialysis.

    N Engl J Med 2001; 344:102-7
13. Auckley D, Schmidt-Nowara W, Brown L. Reversal of sleep apnea hypopnea syndrome in end-stage renal disease after kidney transplantation. Am J Kidney Dis 1999;34:739-744
14. Langevin B, Fougue D, Leger P, Robert D. Sleep apnea syndrome and end-stage renal disease. Cure after renal transplantation. Chest 1993;103:1330-1335
15. Vallance P, Leone A, Calver A, Collier J, Moncada S. Accumulation of an endogenous inhibitor of nitric oxide synthesis in chronic renal failure.

    Lancet. 1992 Mar 7;339(8793):572-5.
16. Kielstein J, Boger R, Bode-Boger S et al. Asymmetric Dimethylarginine Plasma Concentrations Differ in Patients with End-Stage Renal Disease. J Am Soc Nephrol 1999; 10:594-600
17. Kielstein J, Zoccali C. Asymmetric dimethylarginine: a cardiovascular risk factor and a uremic toxin coming of age? Am J Kidney Dis. 2005;46(2):186-202.
18. Saran R, Novak J, Desai A et al. Impact of vitamin E on plasma asymmetric dimethylarginine (ADMA) in chronic kidney disease (CKD): a pilot study.

    Nephrol Dial Transplant. 2003 Nov;18(11):2415-20.
19. Tepel M, van der Giet M, Statz M et al. The antioxidant acetylcysteine reduces cardiovascular events in patients with end-stage renal failure: a randomized, controlled trial. Circulation. 2003 Feb 25;107(7):992-5.
20. Feldman L, Efrati S, Abramsohn R, Yarovoy I, Gersch E, Eviatar E, Averbukh Z, Weissgarten J. N-Acetylcysteine for prevention of gentamicin-induced ototoxicity in hemodialysis patients. J Am Soc Nephrol 2006; 17 (Suppl): 22A
21. Feldman L, Efrati S, Eviatar E, Abramsohn R, Yarovoy I, Gersch E, Averbukh Z, Weissgarten J. N-Acetylcysteine ameliorates gentamicin-induced ototoxicity in hemodialysis patients. Kidney Int 2007 ( in press)

ELIGIBILITY:
Inclusion Criteria:

* The study will include 20 patients with ESRD, treated with chronic hemodialysis in Assaf Harofeh Medical Center and suffering from sleep disturbances, such as frequent arousals, snoring, daytime sleepiness.

Exclusion Criteria:

Patients will be excluded from the study if they are:

* Recently started treated with chronic dialysis: less than 3 months.
* Survived recent major illness, requiring hospitalisation in the last 3 months.
* Patients with acute renal failure
* Currently treated with antioxidants ( NAC, vitamin E ets.)
* Current use of sleep pills

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Leonid S Feldman, MD, Principal Investigator — Assaf Harofeh MC
Locations (1):
- Nephrology Division, Assaf Harofeh Medical Center, Ẕerifin, Israel